CLINICAL TRIAL: NCT02296593
Title: Monitorage Continu du Lactate et de la glycémie Par Microdialyse : Une étude de Validation en Chirurgie Cardiaque.
Brief Title: Continuous MONItoring of Blood LActate and Glucose Levels Using a New Central Veinous Microdialysis Catheter Device
Acronym: MONILAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A14-D36-VOL.22
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Other Functional Disturbances Following Cardiac Surgery
Keywords: lactate; continuous lactate monitoring; continuous blood glucose monitoring; EIRUS; blood glucose; cardiac surgery; central veinous catheter; microdialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for determination of lactate and glucose blood levels
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: comparison of blood lactate and glucose levels — comparison of blood lactate and glucose levels with the reference method (co oxymetry) and a new central veinous catheter microdialysis system provided by MAQUET. (Critical Care AB, Solna, Sweden.)
  Other Names: EIRUS; continuous lactate monitoring; continuous glycemia monitoring; central veinous catheter; microdialysis system; MAQUET

SUMMARY:
Continuous lactate and glucose blood levels

DETAILED DESCRIPTION:
MAQUET Group offers a new device that gives real time blood lactate and glucose levels. It is a new central veinous catheter with a microdialysis system. It is planted in the superior vena cava. It has not yet been used and validated with a clinical purpose, and particularly in cardiac surgery.

For now, reference method for determining blood lactate and glucose levels is co oxymetry.

This new simple device could provide great fluency for determining blood lactate and glucose levels. It could allow medical teams gain time for diagnosis and treatment of both hyperlactatemia and hyperglycemia.

The primary outcome of this study was to compare blood lactate and glucose absolute measures provided with the MAQUET new device (Maquet Critical Care AB, Solna, Sweden) and with co oxymetry.

The secondary outcome of this study was to compare variations of these absolutes measures.

ELIGIBILITY:
Inclusion Criteria:

* Men or women more than 18 years old.
* Cardiac surgery.
* Central veinous catheter in superior vena cava.

Exclusion Criteria:

* Men or women less than 18 years old.
* Pregnant women.
* Central veinous catheter not in superior vena cava.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of cardiac surgery. (planned or for emergencies)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
comparison of absolute blood lactate and glucose levels with the reference method (co oxymetry) and a new method using a device providing real time measures of lactate and glycemia with a central veinous catheter microdialysis system. | 1 day
  Central veinous catheter, EIRUS (Maquet Critical Care AB, Solna, Sweden)

SECONDARY OUTCOMES:
comparison of variations of blood lactate and glycemia levels with the reference method (co oxymetry) and a new method using a device providing real time measures of lactate and glycemia. (EIRUS) with a central veinous catheter microdialysis system. | 1 day
  Central veinous catheter, EIRUS (Maquet Critical Care AB, Solna, Sweden)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, Basse Normandie, France

REFERENCES:
- [Derived] Gouezel C, Lorne E, Bonnet V, Fradin S, Saplacan V, Gerard JL, Hanouz JL, Fellahi JL, Fischer MO; FHT (French Hemodynamic Team). Assessment of changes in lactate concentration with intravascular microdialysis during high-risk cardiac surgery using the trend interchangeability method. Br J Anaesth. 2017 Dec 1;119(6):1110-1117. doi: 10.1093/bja/aex338. PMID 29028910